CLINICAL TRIAL: NCT03840252
Title: Progression of Striatal and Extrastriatal Degeneration in PD and PSP Patients: a Longitudinal Prospective Study for Correlation Between Clinical Manifestations, Gait Analysis and Functional/Diffusion MRI
Brief Title: Progression of Striatal and Extrastriatal Degeneration in PD and PSP Patients
Acronym: PARKONTHEWAY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele Roma (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RP 06/15
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2020-05

CONDITIONS: Parkinson Disease (PD); Paralysis; Supranuclear
Keywords: 3D-gait analysis; Magnetic Resonance Imaging
MeSH Terms: conditions — Parkinson Disease; Paralysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PD patients: Parkinson's disease group (Active Comparator): Diagnosis of idiopathic PD by United Kingdom Brain Bank criteria, exclusion of other significant neurological or orthopedic problems; ages of 21-90; able to walk 25 feet unassisted and without any assistive device.
  Imaging: rsfMRI, diffusion tensor imaging; Motor evaluation: 3D gait analysis; Movement Disorder Society (MDS)-UPDRS Behavioral: PD-MCI-specific Level II battery (Mov Dis. 2015 Mar; 30(3): 402-406)
  Interventions: Diagnostic Test: 3D gait analysis; Diagnostic Test: rsfMRI; Diagnostic Test: Montreal Cognitive assesment (MoCA)
- PSP patients (Active Comparator): Application of the National Institute of Neurological Disorders and Stroke and Society for Progressive Supranuclear Palsy (NINDS-SPSP) criteria for the clinical diagnosis of "probable" PSP, evaluation of PSP rating scale, exclusion of other significant neurological or orthopedic problems; ages of 21-90; able to walk 25 feet unassisted and without any assistive device.
  Imaging: rsfMRI, diffusion tensor imaging; Motor evaluation: 3D gait analysis;MDS-UPDRS Behavioral: PD-MCI-specific Level II battery (Mov Dis. 2015 Mar; 30(3): 402-406)
  Interventions: Diagnostic Test: 3D gait analysis; Diagnostic Test: rsfMRI; Diagnostic Test: Montreal Cognitive assesment (MoCA)
- HC: healthy control group (Active Comparator): Healthy adults ages 21-90 without movement disorders, psychiatric disorders, or dementia.
  Imaging: rsfMRI, diffusion tensor imaging; Motor evaluation: 3D gait analysis; Behavioral: PD-Mild Cognitive Impairment (MCI)-specific Level II battery (Mov Dis. 2015 Mar; 30(3): 402-406)
  Interventions: Diagnostic Test: 3D gait analysis; Diagnostic Test: rsfMRI; Diagnostic Test: Montreal Cognitive assesment (MoCA)

INTERVENTIONS:
Diagnostic Test: 3D gait analysis — Computed analysis of posture and gait pattern and motor performance by kinematic and kinetics parameters analysis such as the step length, gait velocity, stride time variability, 3D joint kinematics, ground reaction forces, joint kinetics
Diagnostic Test: rsfMRI — MR scans acquired by 1.5 Tesla (Siemens Medical Systems, Erlangen, Germany).
  Other Names: resting state functional magnetic resonance (rsfMRI)
Diagnostic Test: Montreal Cognitive assesment (MoCA) — Standard clinical questionnaire

SUMMARY:
This longitudinal study aims to research cognitive and gait phenotypes of Parkinson's disease and Supranuclear Palsy as well as to provide markers to track diseases progression using a multi-modality approach based on 3D-gait analysis and MR Imaging.

Specifically, this study want to identify cognitive pattern and gait-related cerebral diffusion/functional connectivity in PD and PSP patients and to verify their progression over a period of 18 months.

In summary, the current protocol proposed to investigate the following issues:

* to perform a multifactorial quantitative analysis of outcomes for PD and PSP compared to a control group in order to categorize cognitive and gait pattern in the group of patients and verify if the gait can be useful as discriminator for diagnosis.
* to analyze whether diffusion and resting-state functional connectivity indices are correlated with clinical disease severity scores and motor scores and how they change over time (18 months later).

DETAILED DESCRIPTION:
Gait disorder is one of the key features of Parkinson's disease (PD), often leading to loss of mobility and severe disability. Yet in the early stages of disease, examination of gait may lead to inconclusive results for differential diagnosis between PD and other parkinsonism because slow and small stepped walking is often unspecific and can be related to age, depressive mood, or to a presence of neurodegenerative atypical parkinsonism (AP) such as Progressive Supranuclear Palsy (PSP).

At the same time, emerging evidence indicates that early disturbances in cognitive processes such as attention, executive function, and working memory are associated with slower gait and gait instability during single and dual-task testing.

It is therefore crucial to carefully investigate the multiple cognitive domains in order to identify possible mild cognitive deficits in PD and PSP patients and to correlate them with gait disorders.

The use of quantitative movement analysis with 3D-gait analysis allow an objective multifactorial evaluation of the functional limitation related to PD and PSP patients and can be used to analyze the gait in pathologies characterized by gait impairment compared to healthy control (HC).

This longitudinal clinical study aims to analyze cognitive profiles and gait pattern (with 3D-gait analysis) and their progression (18 months later) in a PD- and a PSP-group, respect to HC group.

Moreover, with the Magnetic Resonance Imaging (MRI), the study want to research for possible gait-related cerebral diffusion/functional connectivity alterations and their changes over time.

The specific aims of the project are:

* To perform a multifactorial quantitative analysis of outcomes for PD and PSP compared to a control group in order to categorize the gait in the group of patients and verify if the gait can be useful as discriminator for diagnosis.
* To detect possible cognitive deficits in Parkinson's Disease and PSP more corelated with gait disturbances.
* To analyze whether diffusion and resting-state functional connectivity indices are correlated with clinical disease severity scores and motor scores and how they change over time (18 months later).
* To identify gait-related cerebral diffusion/functional connectivity in PD and PSP patients and to verify their progression over a period of 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic PD by United Kingdom (UK) Brain Bank criteria and PSP according to NINDS-SPSP criteria, without other significant neurological or orthopedic problems;
* ages of 20-80;
* able to walk 25 feet unassisted and without any assistive device

Exclusion Criteria:

* History of epileptic seizures, head injury, other neurological disorders.
* Cardiac pacemaker implantation

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2015-09-23 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Gait profile Score (GPS) in PD and PSP patients | 18 months
  GPS quantifies the gait pattern deviation of the patient respect to normality range

CONTACTS AND LOCATIONS:
Overall Officials: Fabrizio Stocchi, MD, PhD, Study Director — IRCCS San Raffaele Pisana
Locations (1):
- Casa di cura San Raffaele Cassino, Cassino, Frosinone, Italy

IPD SHARING:
Plan to Share IPD: No